CLINICAL TRIAL: NCT06452537
Title: A Randomized, Controlled, Multicenter Study To Evaluate the Safety and Efficacy of Tocilizumab In Patients With Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD)
Brief Title: Safety and Efficacy of Tocilizumab in Patients With Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease
Acronym: TOMATO
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Chao Zhang, Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024035
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease
MeSH Terms: conditions — Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease | interventions — tocilizumab; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab with oral prednisone (Experimental): Tocilizumab will be intravenously administered as the dosage of 8 mg/kg every 4 weeks, with oral prednisone
  Interventions: Drug: Tocilizumab; Drug: Prednisone
- Prednisone (Experimental)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be intravenously administered as the dosage of 8 mg/kg every 4 weeks, with oral prednisone.
  Other Names: ACTEMRA®
  Arms: Tocilizumab with oral prednisone
Drug: Prednisone — Prednisone tapering protocol : If the starting dose is over 20mg/day, then reduce by one tablet weekly. Until the dose is reduced to 20mg/day then 20mg/day for two weeks→17.5mg/day for two weeks→12.5mg for four weeks→10mg for four weeks→7.5mg as a maintain dosage

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Tocilizumab in MOGAD.

DETAILED DESCRIPTION:
Myelin oligodendrocyte glycoprotein antibody-associated disease (MOGAD) is a rare autoimmune disease of the central nervous system, which can cause optic neuritis, myelitis, brainstem encephalitis, or encephalitis. The specific autoantibody against myelin oligodendrocyte glycoprotein antibody (MOG-IgG) has been indicated to contribute to the pathogenesis of the disease. Data from several cohorts suggests that around 50% of adult patients with MOG-IgG may relapse within the first two years of the disease, with most of relapses occurring early after disease onset. Few randomized controlled trials have ever been performed and therapeutic guidelines for this disease remain unclear especially after a single event. There is no drug approved for MOGAD by FDA. IL-6 is a pro-inflammatory cytokine which can promotes B cell activation, blood-brain barrier dysfunction, leukocyte migration, and the production of autoantibodies. Tocilizumab (ACTEMRA®), a humanized monoclonal antibody against the IL-6 receptor, has shown beneficial clinical effects and reduction of the risk of relapses in some patients with MOGAD. However, the efficacy of tocilizumab in MOGAD warrants further clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are aged ≥12 years at the time of signing Informed Consent Form
2. Confirmed diagnosis of MOGAD with a history of ≥1 MOGAD relapse in the 12 months prior to screening or ≥2 attacks in the 24 months prior to screening
3. Anti-MOG antibody seropositive
4. For women of childbearing potential: participants who agree to remain abstinent or use adequate contraception during the treatment period and for at least 3 months after the final dose of tocilizumab
5. Patients must give written informed consent

Exclusion Criteria:

1. Any concomitant disease other than MOGAD that may require treatment with oral immunosuppressants or prednisone at doses >20 mg/day (or equivalent)
2. Receipt of the following at any time prior to randomization Alemtuzumab Total lymphoid irradiation Bone marrow transplant T-cell vaccination therapy Receipt of rituximab or any experimental B-cell depleting agent within 6 months prior screening and B-cells below the lower limit of normal.

   Receipt of intravenous immunoglobulin (IVIG) or plasma exchange (PE) within 1 month prior to randomization.

   Receipt of any of the following within 3 months prior to randomization:

   Natalizumab (Tysabri®). Methotrexate Mitoxantrone Cyclophosphamide Eculizumab

   Receipt of any of the following within 6 weeks prior to randomization:

   Tacrolimus Cyclosporin Mycophenolate mofetil
3. Participants who are pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of tocilizumab
4. Participants with active or presence of recurrent bacterial, viral, fungal, mycobacterial infection, or other infection at baseline
5. Participants with evidence of latent or active tuberculosis (excluding patients receiving chemoprophylaxis for latent tuberculosis infection)
6. Participants with positive screening tests for hepatitis B and C
7. Receipt of live or live attenuated vaccine within 6 weeks prior to baseline
8. Known history of a severe allergy or reaction to any biologic therapy.
9. History of alcohol, drug, or chemical abuse, or a recent history of such abuse < 1 year prior to randomization
10. WBC < 3.0 × 10^3/mL, ANC < 2.0 × 10^3/mL, PLT < 10 × 10^4/mL, AST or ALT>1.5 ×ULN, Lymphocyte count < 0.5 × 10^3/mL

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Time from randomization to the first MOGAD relapse as determined by an adjudication committee | Baseline, Up To 60 Weeks (End of Study)
  An adjudicated relapse was defined by the protocol and positively adjudicated by the relapse adjudication committee.

SECONDARY OUTCOMES:
Percentage of Participants With Worsening in Expanded Disability Severity Scale (EDSS) Score From Baseline to the end of study | Baseline, Up To 60 Weeks (End of Study)
  Disease-related disability was measured by the EDSS. The EDSS was an ordinal clinical rating scale that ranges from 0 (normal neurologic examination) to 10 (death) in half-point increments. A decrease in score indicates improvement
Dosage of oral steroid at the end of the TOMATO trial | Baseline, Up To 60 Weeks (End of Study)
  Dosage of oral steroid at the end of the TOMATO trial
Sera MOG-IgG Concentration Over Time | Baseline, Weeks 12, 24, 36, 48, 60 Weeks (End of Study)
  Sera MOG-IgG Concentration was measured by Cell-Based Assay (CBA)
Number of Participants With Adverse Events (AEs) | Baseline, Up To 60 Weeks (End of Study)
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship
Number of Participants With Adverse Events Serious Adverse Events (SAEs) | Baseline, Up To 60 Weeks (End of Study)
  A SAE was any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization
Number of the lesion of the MRI T2WI | Baseline, Weeks 12, 24, 36, 48, 60 Weeks (End of Study)
  Number of the lesion of the MRI T2WI

CONTACTS AND LOCATIONS:
Overall Officials: Chao Zhang, M.D., Ph.D, Principal Investigator — Tianjin Medical University General Hospital
Locations (22):
- China (22):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Hebei Children's Hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou, Henan
  - Ordos Central Hospital, Ordos, Inner Mongolia
  - The Third Affiliated Hospital of Soochow University, Changzhou, Jiangsu
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang Uygur Autonomous Region
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The First Affiliated Hospital of Tsinghua University, Beijing
  - XuanWu Hospital Capital Medical University, Beijing
  - Huashan Hospital, Fudan University, Shanghai
  - Tianjin Huanhu Hospital, Tianjin
  - Tianjin Children's Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No